CLINICAL TRIAL: NCT04252742
Title: Comprehensive Assessment of Erenumab Efficacy in Subjects With High Frequency Episodic Migraine With at Least 1 Previously Failed Preventive Treatment: a Global, Double-blind, Placebo-controlled Phase 4 Study
Brief Title: Erenumab - Comprehensive Assessment of Efficacy in (High-Frequency) Episodic Migraine
Acronym: EMBRACE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20190008; 2019-003646-33 (EudraCT Number)
Record Dates: First submitted 2020-01-22; First posted 2020-02-05 (Actual); Results first posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-07

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — erenumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Erenumab (Experimental): The 4-month DBTP has 2 phases:
  * Main double-blind treatment phase (M-DBTP, months 1 to 3) that will assess the effect of erenumab on metrics such as time spent in at least moderate pain, peak migraine severity, and functional impairment.
  * Exploratory DBTP (E-DBTP, month 4) that will assess the impact of erenumab on the acute response to treatment with oral triptan therapy as well as non-ictal burden.
  Interventions: Drug: Erenumab
- Placebo (Experimental): The 4-month DBTP has 2 phases:
  * Main DBTP (M-DBTP, months 1 to 3) that will assess the effect of erenumab on metrics such as time spent in at least moderate pain, peak migraine severity, and functional impairment.
  * Exploratory DBTP (E-DBTP, month 4) that will assess the impact of erenumab on the acute response to treatment with oral triptan therapy as well as non-ictal burden.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Erenumab — 140 mg, 2 consecutive injections of 70 mg
  Arms: Erenumab
Drug: Placebo — 2 consecutive injections
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the treatment benefit of erenumab on headache duration of at least moderate pain intensity.

ELIGIBILITY:
Key inclusion criteria include:

* Age greater than or equal to 18 years upon entry into initial screening.
* Documented history of migraine with or without aura according to the International Headache Society (IHS) International Classification of Headache Disorders, Third Edition (ICHD-III) for greater than or equal to 12 months.
* Have high-frequency episodic migraine (HFEM): Defined as history of ≥ 7 to < 15 migraine days and < 15 headache days per month on average during the 3 months prior to screening.
* History of ≥ 4 migraine attacks of at least moderate severity per month on average during the 3 months prior to screening.
* History of treatment failure with at least 1 preventive treatment for migraine. Failure of preventive treatment for migraine is defined as treatment discontinuation due to lack of efficacy, adverse event, or general poor tolerability.
* Regular use of an oral triptan (using only eletriptan, rizatriptan, sumatriptan, or zolmitriptan) for acute migraine treatment, and typically initiating acute treatment with an oral triptan on > 50% of attacks of at least moderate pain intensity. Regular use is defined as ≥ 4 days of oral triptan use per month during the 3 months prior to screening.

Key exclusion criteria include:

* History of hemiplegic migraine, cluster headache, or other trigeminal autonomic cephalalgia.
* Has any medical contraindication to the use of an oral triptan.
* Previously treated with erenumab.
* Previously treated with a gepant (small molecule calcitonin gene related peptide receptor [CGRP-R] antagonist) in a preventive fashion in a manner consistent with migraine prevention that either:

  1. In the opinion of the investigator, did not offer any evidence of a therapeutic response or
  2. Was discontinued for less than 12 weeks from the date of initial screening or
  3. Was previously discontinued due to a known adverse drug reaction
* Currently being treated with lasmiditan and/or a gepant in the acute setting.
* No therapeutic response with greater than 4 of the defined medication categories after an adequate therapeutic trial.
* Currently has a history of consistent excellent response to oral triptans, defined as achievement of pain-freedom in ≤ 1 hour for ≥ 50% of treated attacks of at least moderate pain intensity during the 3 months prior to screening.
* Use of triptans administered via a non-oral (e.g. subcutaneous [SC] or intranasal delivery systems) or sublingual route at the time of screening, during the run-in and baseline periods, and throughout the study duration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 512 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2023-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (91):
- United States (31):
  - Long Beach Clinical Trials Services Inc, Long Beach, California
  - Clinical Research Institute, LLC, Los Angeles, California
  - Mountain Neurological Research Center, Basalt, Colorado
  - Denver Neurological Clinic, Denver, Colorado
  - Summit Headache and Neurologic Institute, Englewood, Colorado
  - JEM Research Institute, Atlantis, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Visionary Investigators Network, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Heuer Medical Doctor Research LLC, Orlando, Florida
  - Neurology Associates of Ormond Beach, Ormond Beach, Florida
  - Visionary Investigators Network, Pembroke Pines, Florida
  - Saint Lukes Clinic, Meridian, Idaho
  - Chicago Headache Center and Research Institute, Chicago, Illinois
  - Boston Clinical Trials, Boston, Massachusetts
  - New England Regional Headache Center Inc, Worcester, Massachusetts
  - Michigan Head Pain and Neurological Institute, Ann Arbor, Michigan
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Clinvest Research LLC, Springfield, Missouri
  - Mercy Health Research, St Louis, Missouri
  - Papillion Research Center, Papillion, Nebraska
  - Forte Family Practice, Las Vegas, Nevada
  - Dent Neurosciences Research Center, Amherst, New York
  - American Clinical Research Institute LLC, Beavercreek, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Summit Research Network, Portland, Oregon
  - Palmetto Clinical Trial Services, Greenville, South Carolina
  - Nashville Neuroscience Group, Nashville, Tennessee
  - FutureSearch Trials of Neurology, Austin, Texas
  - North Texas Institute of Neurology and Headache, Frisco, Texas
- Bulgaria (7):
  - University Multiprofile Hospital for Active Treatment - Dr Georgi Stranski EAD, Pleven
  - University Multiprofile Hospital for Active Treatment Sveti Georgi EAD, Plovdiv
  - Multiprofile Hospital for Active Treatment in neurology and psychiatry Sveti Naum EAD, Sofia
  - University First Multiprofile Hospital for Active Treatment - Sofia Sveti Yoan Krastitel EAD, Sofia
  - Medical Center Excelsior OOD, Sofia
  - University Multiprofile Hospital for Active Treatment Alexandrovska EAD, Sofia
  - Medical Center New Rehabilitation Center EOOD, Stara Zagora
- Czechia (8):
  - Neurologie Brno sro, Brno
  - Fakultni nemocnice u svate Anny v Brne, Brno
  - Poliklinika Chocen, Neurohk sro, Choceň
  - Brain-soultherapy sro, Kladno
  - Dado Medical sro, Prague
  - FORBELI sro, Prague
  - Institut Neuropsychiatricke pece, Prague
  - NeuroMed Zlin sro, Zlín
- Hungary (6):
  - Obudai Egeszsegugyi Centrum Kft, Budapest
  - High Tech Medical Kft, Budapest
  - Uno Medical Trials Kft, Budapest
  - S-Medicon Kutatasi Centrum, Budapest
  - Orszagos Mentalis, Ideggyogyaszati es Idegsebeszeti Intezet, Budapest
  - Obudai Egeszsegugyi Centrum Kft, Zalaegerszeg
- Italy (10):
  - Ospedale Bellaria Carlo Alberto Pizzardi, Bologna
  - Azienda Socio Sanitaria Teritoriale Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliera Universitaria Renato Dulbecco, Catanzaro
  - Ospedale Policlinico San Martino IRCCS, Genoa
  - IRCCS Ospedale San Raffaele, Milan
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan
  - Fondazione Istituto Neurologico Nazionale C Mondino IRCCS, Pavia
  - Policlinico Universitario Campus Biomedico, Roma
  - IRCCS San Raffaele Pisana, Roma
  - Azienda della scienza di Torino, Torino
- Poland (14):
  - Centrum Badan Klinicznych PI-House Spzoo, Gdansk
  - Gabinet Diagnostyki i Leczenia Osteoporozy Prof Wojciech Pluskiewicz, Gliwice
  - Care Clinic Spzoo Care Clinic Centrum Medyczne, Katowice
  - Vita Longa Spzoo, Katowice
  - NZOZ Neuromed M i M Nastaj Spolka Partnerska, Kraśnik
  - AppleTreeClinics Network Spzoo, Lodz
  - M-Zdrowie, Lodz
  - NZOZ Neuromed M i M Nastaj Spolka Partnerska, Lublin
  - Instytut Zdrowia Dr Boczarska-Jedynak Spzoo SpKom, Oświęcim
  - Osrodek Badan Klinicznych Cromed, Poznan
  - Prywatny Gabinet Neurologiczny Iwona Rosciszewska-Zukowska, Rzeszów
  - Migre Polskie Centrum Leczenia Migreny Anna Gryglas-Dworak, Wroclaw
  - Centrum Medyczne Oporow, Wroclaw
  - Vistamed and Vertigo Sp z o o, Wroclaw
- Portugal (4):
  - Hospital da Luz, SA, Lisbon
  - Centro Hospitalar Universitario de Lisboa Norte, EPE - Hospital de Santa Maria, Lisbon
  - Hospital Cuf Sintra, Sintra
  - Campus Neurologico Senior, Torres Vedras
- Romania (3):
  - Spitalul Universitar de Urgenta Militar Central Dr. Carol Davila, Bucharest
  - Spitalul Universitar de Urgenta Bucuresti, Bucharest
  - Spitalul Clinic Judetean de Urgenta Pius Brinzeu Timisoara, Timișoara
- Spain (8):
  - Hospital Universitario Virgen del Rocio, Seville, Andalusia
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza, Aragon
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Clinico Universitario de Valladolid, Valladolid, Castille and León
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Clinico Universitario de Valencia, Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s)and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 61 study centers in North America and Europe from September 2020 to October 2023.
Pre-assignment Details: Eligible adult participants with high frequency episodic migraine (EP) who met specific eligibility criteria during a 2-week run-in period and 4-week baseline period entered the double-blind treatment period (DBTP). The DBTP included a 12-week main-DBTP (M-DBTP) and a 4-week exploratory DBTP (E-DBTP)
Groups:
- Placebo: Participants were randomized to receive matching placebo subcutaneously (SC) every 4 weeks (Q4W) for up to 16 weeks.
- Erenumab 140 mg SC Q4W: Participants were randomized to receive 140 mg erenumab SC Q4W for up to 16 weeks in the DBTP.
Period: Overall Study
Arm/Group | Placebo | Erenumab 140 mg SC Q4W
Started | 256 | 256
Received Investigational Product (IP) | 256 | 254
Completed | 241 | 244
Not Completed | 15 | 12
Not completed — Decision by sponsor | 0 | 2
Not completed — Withdrawal by Subject | 15 | 9
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set included all participants who were randomized in the study.
Groups:
- Placebo: Participants were randomized to receive matching placebo SC QW4 for up to 16 weeks in the DBTP.
- Total: Total of all reporting groups
Arm/Group | Placebo | Erenumab 140 mg SC Q4W | Total
Number analyzed (Participants) | 256 | 256 | 512
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (10.2) | 41.9 (10.9) | 42.2 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 222 | 220 | 442
  Male | 34 | 36 | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 7 | 14
  Not Hispanic or Latino | 248 | 249 | 497
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 253 | 252 | 505
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Monthly Hours of at Least Moderate Headache Pain Intensity [Mean (Standard Deviation); unit: hours/month] — At least moderate headache pain intensity was defined as headache pain intensity reported as 'Moderate' or 'Severe' based on the 3-level headache pain intensity scale. Worst or peak pain intensity during a headache was collected using the e-diary in 3-levels (mild, moderate or severe). The duration of headaches with at least moderate pain intensity was collected. Baseline data was collected during the 4-week baseline period. Population: Participants with observed data within the 4-week baseline period are included.
  hours/month
    number analyzed (Participants) | 255 | 256 | 511
    (all) | 47.382 (29.302) | 48.843 (29.502) | 48.114 (29.383)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Monthly Hours of at Least Moderate Headache Pain Intensity Over Months 1, 2, and 3
Description: At least moderate headache pain intensity was defined as headache pain intensity reported as 'Moderate' or 'Severe' based on the 3-level headache pain intensity scale. Worst or peak pain intensity during a headache was collected using the e-diary in 3-levels (mild, moderate or severe). The duration of headaches with at least moderate pain intensity was collected. A negative change from baseline indicates a reduction in mean monthly hours of at least moderate headache pain intensity. Change from baseline in mean monthly measurement is the arithmetic mean of the monthly change from baseline values for the months considered with observed data, if there was at least one observed monthly value.
  The least squares mean (LSM) estimates of change from baseline in reported headache pain intensity utilized a linear mixed model which included treatment, visit, treatment-by-visit interaction, and baseline value as covariates and assumed a first-order auto regression covariance structure.
Time Frame: Baseline, Month 1, Month 2, and Month 3
Population: The M-DBTP efficacy analysis set consisted of a subset the full analysis set (all participants randomized in the study) who received at least 1 dose of IP and had observed monthly hours of at least moderate headache pain intensity at baseline and at least 1 measurement during the M-DBTP.
Measure: Least Squares Mean (Standard Error); unit: hours/month
Arm/Group | Placebo | Erenumab 140 mg SC Q4W
Number analyzed (Participants) | 251 | 253
hours/month | -23.38 (1.26) | -31.33 (1.25)
Statistical Analysis 1: Comparison: Placebo vs Erenumab 140 mg SC Q4W; Test type: Superiority; p < 0.001, Mixed Models Analysis — Nominal p-value is presented without multiplicity adjustment; Treatment, visit, treatment-by-visit interaction, and baseline value as covariates; LSM difference = -7.95, 95% CI 2-sided [-11.45 to -4.46] — Erenumab 140 mg SC Q4W - Placebo

2. Secondary Outcome: Change From Baseline in Mean Monthly Physical Function Domain Score as Measured by the Migraine Functional Impact Questionnaire (MFIQ) Over Months 1, 2, and 3
Description: The MFIQ is a self-administered 26-item instrument measuring the impact of migraine on broader functioning including on Physical Functioning (5 items). Participants responded to items using a 5-point scale assigned scores from 1 to 5, with 5 representing the greatest burden. Each domain score was calculated as the sum of the item responses and rescaled to a 0 to 100 scale, with higher scores representing greater burden. The recall period was the past 7 days. A negative change from baseline indicates an improvement in burden. Change from baseline in mean monthly scores is the arithmetic mean of the monthly change from baseline values for the months considered with observed data, if there was at least one observed monthly value.
  The LSM estimates utilized a linear mixed model which included treatment, visit, treatment-by-visit interaction, and baseline value as covariates and assumed a first-order auto regression covariance structure.
Time Frame: Baseline, Month 1, Month 2, and Month 3
Population: The M-DBTP efficacy analysis set consisted of a subset the full analysis set (all participants randomized in the study) who received at least 1 dose of IP and had observed monthly hours of at least moderate headache pain intensity at baseline and at least 1 measurement during the M-DBTP. Data for participants included in the model for the MFIQ Physical Function Domain are presented.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Erenumab 140 mg SC Q4W
Number analyzed (Participants) | 239 | 244
score on a scale | -22.92 (1.25) | -30.28 (1.23)
Statistical Analysis 1: Comparison: Placebo vs Erenumab 140 mg SC Q4W; Test type: Superiority; p < 0.001, Mixed Models Analysis — Nominal p-value is presented without multiplicity adjustment; Treatment, visit, treatment-by-visit interaction, and baseline value as covariates; LSM difference = -7.36, 95% CI 2-sided [-10.80 to -3.92] — Erenumab 140 mg SC Q4W - Placebo

3. Secondary Outcome: Change From Baseline in Mean Monthly Usual Activities Domain Score as Measured by the MFIQ Over Months 1, 2, and 3
Description: The MFIQ is a self-administered 26-item instrument measuring the impact of migraine on broader functioning including Impact on Usual Activities (10 items). Participants responded to items using a 5-point scale assigned scores from 1 to 5, with 5 representing the greatest burden. Each domain score was calculated as the sum of the item responses and rescaled to a 0 to 100 scale, with higher scores representing greater burden. The recall period was the previous 7 days. A negative change from baseline indicates an improvement in burden. Change from baseline in mean monthly scores is the arithmetic mean of the monthly change from baseline values for the months considered with observed data, if there was at least one observed monthly value.
  The LSM estimates utilized a linear mixed model which included treatment, visit, treatment-by-visit interaction, and baseline value as covariates and assumed a first-order auto regression covariance structure.
Time Frame: Baseline, Month 1, Month 2, and Month 3
Population: The M-DBTP efficacy analysis set consisted of a subset the full analysis set (all participants randomized in the study) who received at least 1 dose of IP and had observed monthly hours of at least moderate headache pain intensity at baseline and at least 1 measurement during the M-DBTP. Data for participants included in the model for the MFIQ Usual Activities Domain are presented.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Erenumab 140 mg SC Q4W
Number analyzed (Participants) | 239 | 244
score on a scale | -23.98 (1.17) | -31.08 (1.16)
Statistical Analysis 1: Comparison: Placebo vs Erenumab 140 mg SC Q4W; Test type: Superiority; p < 0.001, Mixed Models Analysis — Nominal p-value is presented without multiplicity adjustment; Treatment, visit, treatment-by-visit interaction, and baseline value as covariates; LSM difference = -7.10, 95% CI 2-sided [-10.34 to -3.87] — Erenumab 140 mg SC Q4W - Placebo

4. Secondary Outcome: Change From Baseline in Mean Monthly Emotional Functioning Domain Score as Measured by the MFIQ Over Months 1, 2, and 3
Description: The MFIQ is a self-administered 26-item instrument measuring the impact of migraine on broader functioning including Impact on Emotional Functioning (5 items). Participants responded to items using a 5-point scale assigned scores from 1 to 5, with 5 representing the greatest burden. Each domain score was calculated as the sum of the item responses and rescaled to a 0 to 100 scale, with higher scores representing greater burden. The recall period was the previous 7 days. A negative change from baseline indicates an improvement in burden. Change from baseline in mean monthly scores is the arithmetic mean of the monthly change from baseline values for the months considered with observed data, if there was at least one observed monthly value.
  The LSM estimates utilized a linear mixed model which included treatment, visit, treatment-by-visit interaction, and baseline value as covariates and assumed a first-order auto regression covariance structure.
Time Frame: Baseline, Month 1, Month 2, and Month 3
Population: The M-DBTP efficacy analysis set consisted of a subset the full analysis set (all participants randomized in the study) who received at least 1 dose of IP and had observed monthly hours of at least moderate headache pain intensity at baseline and at least 1 measurement during the M-DBTP. Data for participants included in the model for the MFIQ Emotional Functioning Domain are presented.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Erenumab 140 mg SC Q4W
Number analyzed (Participants) | 239 | 244
score on a scale | -22.77 (1.34) | -29.83 (1.33)
Statistical Analysis 1: Comparison: Placebo vs Erenumab 140 mg SC Q4W; Test type: Superiority; p < 0.001, Mixed Models Analysis — Nominal p-value is presented without multiplicity adjustment; Treatment, visit, treatment-by-visit interaction, and baseline value as covariates; LSM difference = -7.05, 95% CI 2-sided [-10.76 to -3.34] — Erenumab 140 mg SC Q4W - Placebo

5. Secondary Outcome: Change From Baseline in Mean Monthly Social Functioning Domain Score as Measured by the MFIQ Over Months 1, 2, and 3
Description: The MFIQ is a self-administered 26-item instrument measuring the impact of migraine on broader functioning including Impact on Social Functioning (5 items). Participants responded to items using a 5-point scale assigned scores from 1 to 5, with 5 representing the greatest burden. Each domain score was calculated as the sum of the item responses and rescaled to a 0 to 100 scale, with higher scores representing greater burden. The recall period was the previous 7 days. A negative change from baseline indicates an improvement in burden. Change from baseline in mean monthly scores is the arithmetic mean of the monthly change from baseline values for the months considered with observed data, if there was at least one observed monthly value.
  The LSM estimates utilized a linear mixed model which included treatment, visit, treatment-by-visit interaction, and baseline value as covariates and assumed a first-order auto regression covariance structure.
Time Frame: Baseline, Month 1, Month 2, and Month 3
Population: The M-DBTP efficacy analysis set consisted of a subset the full analysis set (all participants randomized in the study) who received at least 1 dose of IP and had observed monthly hours of at least moderate headache pain intensity at baseline and at least 1 measurement during the M-DBTP. Data for participants included in the model for the MFIQ Social Functioning Domain are presented.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Erenumab 140 mg SC Q4W
Number analyzed (Participants) | 239 | 244
score on a scale | -25.05 (1.28) | -31.87 (1.27)
Statistical Analysis 1: Comparison: Placebo vs Erenumab 140 mg SC Q4W; Test type: Superiority; p < 0.001, Mixed Models Analysis — Nominal p-value is presented without multiplicity adjustment; Treatment, visit, treatment-by-visit interaction, and baseline value as covariates; LSM difference = -6.82, 95% CI 2-sided [-10.37 to -3.27] — Erenumab 140 mg SC Q4W - Placebo

6. Secondary Outcome: Change From Baseline in Mean Monthly Average Duration of at Least Moderate Headache Pain Intensity in Migraine Attacks Occurring Over Months 1, 2, and 3
Description: At least moderate headache pain intensity was defined as headache pain intensity reported as 'Moderate' or 'Severe' based on the 3-level headache pain intensity scale. Worst or peak pain intensity during a headache was collected using the e-diary in 3-levels (mild, moderate or severe). The duration of headaches with at least moderate pain intensity during a migraine attack was collected. A negative change from baseline indicates a reduction in mean monthly average duration of at least moderate headache pain intensity during a migraine attack. Change from baseline in mean monthly measurement is the arithmetic mean of the monthly change from baseline values for the months considered with observed data, if there was at least one observed monthly value.
  The LSM estimates utilized a linear mixed model which included treatment, visit, treatment-by-visit interaction, and baseline value as covariates and assumed a first-order auto regression covariance structure.
Time Frame: Baseline, Month 1, Month 2, and Month 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Erenumab 140 mg SC Q4W
Number analyzed (Participants) | 251 | 253
hours | -2.78 (0.31) | -3.86 (0.30)
Statistical Analysis 1: Comparison: Placebo vs Erenumab 140 mg SC Q4W; Test type: Superiority; p = 0.013, Mixed Models Analysis — Nominal p-value is presented without multiplicity adjustment; Treatment, visit, treatment-by-visit interaction, and baseline value as covariates; LSM difference = -1.07, 95% CI 2-sided [-1.92 to -0.22] — Erenumab 140 mg SC Q4W - Placebo

7. Secondary Outcome: Change From Baseline in Mean Monthly Average Peak Migraine Pain Intensity as Assessed by the 11-point Numeric Rating Scale (NRS) Over Months 1, 2, and 3
Description: The NRS assesses headache pain intensity ranging from 0 to 10 with a higher score indicating more severe pain. Participants recorded the pain intensity using the e-diary at the headache end-time or in an evening diary entry on a daily basis for an ongoing headache. A negative change from baseline indicates an improvement in pain intensity. Change from baseline in mean monthly scores is the arithmetic mean of the monthly change from baseline values for the months considered with observed data, if there was at least one observed monthly value.
  The LSM estimates utilized a linear mixed model which included treatment, visit, treatment-by-visit interaction, and baseline value as covariates and assumed a first-order auto regression covariance structure.
Time Frame: Baseline, Month 1, Month 2, and Month 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Erenumab 140 mg SC Q4W
Number analyzed (Participants) | 251 | 253
score on a scale | -1.48 (0.13) | -1.96 (0.13)
Statistical Analysis 1: Comparison: Placebo vs Erenumab 140 mg SC Q4W; Test type: Superiority; p = 0.011, Mixed Models Analysis — Nominal p-value is presented without multiplicity adjustment; Treatment, visit, treatment-by-visit interaction, and baseline value as covariates; LSM difference = -0.48, 95% CI 2-sided [-0.85 to -0.11] — Erenumab 140 mg SC Q4W - Placebo

ADVERSE EVENTS:
Time Frame: Day 1 to end of the DBTP (up to 16 weeks)
Description: All-cause mortality is reported for all participants enrolled/randomized in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Arm/Group | Placebo | Erenumab 140 mg SC Q4W
All-Cause Mortality (participants affected / at risk) | 0/256 | 0/256
Serious Adverse Events (participants affected / at risk) | 2/256 | 0/254
Other Adverse Events (participants affected / at risk) | 0/256 | 0/254
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=256) | Erenumab 140 mg SC Q4W (N=254)
COVID-19 pneumonia (Infections and infestations) | 1 | 0
Psychogenic tremor (Psychiatric disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2022-06-29): https://cdn.clinicaltrials.gov/large-docs/42/NCT04252742/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-15): https://cdn.clinicaltrials.gov/large-docs/42/NCT04252742/SAP_001.pdf